CLINICAL TRIAL: NCT06524492
Title: Measurements of Flow in Functional Cerebrospinal Fluid Shunts and Off-Shunt Locations with a Second-Generation Wireless Thermal Anisotropy Measurement Device
Brief Title: Flow Measurements in Functional CSF Shunts and Off-Shunt Locations with a Second-Generation Thermal Device
Status: Completed | Type: Observational
Sponsor: Rhaeos, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-04
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- FlowSense: This study compares the performance of two generations of non-invasive cerebrospinal fluid (CSF) shunt flow assessment devices. Measurements of functional implanted shunts and off-shunt locations will assess the diagnostic non-inferiority of the second-generation device to the first-generation device.
  Interventions: Device: FlowSense

INTERVENTIONS:
Device: FlowSense — This study compares the performance of two generations of non-invasive cerebrospinal fluid (CSF) shunt flow assessment devices. Measurements of functional implanted shunts and off-shunt locations will assess the diagnostic non-inferiority of the second-generation device to the first-generation device.

SUMMARY:
This study compares the performance of two generations of non-invasive cerebrospinal fluid (CSF) shunt flow assessment devices. Measurements of functional implanted shunts and off-shunt locations will assess the diagnostic non-inferiority of the second-generation device to the first-generation device.

ELIGIBILITY:
Inclusion criteria

1. A ventricular CSF shunt with a region of overlying intact skin appropriate in size for application of the study device
2. Signed informed consent by subject or a parent, legal guardian, health care agent, or surrogate decision maker (according to local statutes)
3. Signed medical records release by subject or a parent, legal guardian, health care agent, or surrogate decision maker (according to local statutes)
4. Verbal assent by minors 7 years of age and older who are able to understand the study and communicate their decision

Exclusion criteria

1. Presence of an interfering open wound or edema in the study device measurement area
2. Patient-reported history of serious adverse skin reactions to silicone-based adhesives
3. Previous participation in a Rhaeos clinical study in which FlowSense device measurement data were acquired
4. Patient or caregiver report of new or worsening symptoms of a possible shunt malfunction in the prior 7 days
5. Participation in any other investigational procedural, pharmaceutical, and/or device study that may influence the collection of valid data under this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult patients with an existing ventricular shunt will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2024-07-27 (Actual); Study Completion 2024-07-27 (Actual)

PRIMARY OUTCOMES:
Study Device Sensitivity | Approximately 1 hour
  Study device sensitivity will be calculated as TP / (TP + FN).
Study Device Specificity | Approximately 1 hour
  Study device specificity will be calculated as TN / (TN + FP)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Tampa Marriott Water Street, Tampa, Florida
  - Rhaeos, Inc., Chicago, Illinois
  - Northwest Special Recreation Association, Rolling Meadows, Illinois

IPD SHARING:
Plan to Share IPD: No